CLINICAL TRIAL: NCT06707753
Title: An Open-label, Nonrandomized, Single-arm, Single Dose, Dose-escalation Phase I/IIa Study to Evaluate the Safety and Tolerability of AL-001 Ophthalmic Injection in Subjects with Wet Age-related Macular Degeneration (wAMD)
Brief Title: Safety and Tolerability of AL-001 Ophthalmic Injection in Subjects with WAMD
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Anlong Biopharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AL-001-01
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-02

CONDITIONS: Wet Age-related Macular Degeneration (wAMD)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- AL-001 Dose 1 (Experimental): Injection of low dose
  Interventions: Drug: AL-001
- AL-001 Dose 2 (Experimental): Injection of medium dose
  Interventions: Drug: AL-001
- AL-001 Dose 3 (Experimental): Injection of high dose
  Interventions: Drug: AL-001

INTERVENTIONS:
Drug: AL-001 — Administered via suprachoroidal space injection.

SUMMARY:
This Phase I/IIa study is designed to evaluate the safety, tolerability, preliminary pharmacodynamics and pharmacokinetics in patients with wet age-related macular degeneration. Eligible patients, who meet the inclusion/exclusion criteria and have shown an anatomic response to an anti-VEGF (Vascular Endothelial Growth Factor) injection, will receive a single dose of AL-001 administered via suprachoroidal space injection.

ELIGIBILITY:
Inclusion Criteria:

1. Age≥ 50 and ≤ 80.
2. The study eye was diagnosed with subfoveal active choroidal neovascularization (CNV) lesions secondary to wAMD.
3. Best Corrected Visual Acuity (BCVA) of study eye during screening, Early Treatment of Diabetic Retinopathy Study (ETDRS) letters≤73 and ≥19.
4. The subject or their legal representative agrees to participate in this study and signs a written ICF.

Exclusion Criteria:

1. Non-wAMD induced CNV or macular edema in the study eye.
2. Non-wAMD induced eye conditions that may affect central vision or medical history that may seriously affect central vision in the study eye.
3. Uncontrolled glaucoma in the study eye.
4. History of vitreoretinal surgery, antiglaucoma trabeculectomy, or other anti-glaucoma filtering surgery in the study eye.
5. Refractive interstitial opacity that significantly affects visual function assessment or fundus examination in the study eye.
6. Ametropia (high myopia or high hyperopia) > 8.0D in the study eye, or significant posterior scleral staphyloma in the study eye.
7. Malignant tumor in any eye, including but not limited to eye lymphoma or choroidal melanoma.
8. None of intraocular inflammation in the study eye.
9. Other conditions that may affect compliance or may not be suitable to participate in this trial in the opinion of investigator.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-09-11 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | Week 24
  Incidence of adverse events (AEs) and serious adverse events (SAEs)

SECONDARY OUTCOMES:
Evaluate the effect of AL-001 on BCVA | Week 52
  Mean change from baseline in BCVA

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese Academy of Medical Sciences & Peking Union Hospital, Beijing, China